CLINICAL TRIAL: NCT02609321
Title: Efficacy of Thoracic Paravertebral Block vs Local Anesthesia of the Surgical Wound in Reduction of Acute Post-surgical Pain in Patients With Breast Cancer. Controlled Phase III, Randomized, Single-blind, Superiority Clinical Trial.
Brief Title: Efficacy of Thoracic Paravertebral Block in the Reduction of Acute Post-surgical Pain in Patients With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Cancerología S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDC0001
Record Dates: First submitted 2015-09-14; First posted 2015-11-20 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: Paravertebral; Single injection; Breast surgery; Analgesia
MeSH Terms: conditions — Breast Neoplasms; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic Paravertebral Block (Experimental): to identify the thoracic T3, a parallel line 2.5 cm from the spinous process is drawn and in this place the ultrasound sensor is placed. Ultrasonograph image identifies the transverse process, the intercostal cost-transverse ligament, the pleura and lung. We proceed to insert a needle between the two corresponding transverse processes and positions after passing the cost-ligament posterior intercostal and transverse to the parietal pleura. After negative aspiration for blood, 0.5% bupivacaine anesthetic is administered at doses of 1.5 mg/kg slowly. The volume is defined by the anesthesiologist. The injection of anesthetic is displayed, as well as confirmation of the correct location of the needle because the volume injected above pushes the pleura.
  Interventions: Procedure: Thoracic Paravertebral Block
- Surgical Wound Infiltration (Active Comparator): before the close of the skin, it proceeds to infiltrate the subcutaneous tissue and skin with 0.5% bupivacaine at doses of 1.5 mg/kg, generating the widest possible dissemination of the bupivacaine in the surgical area.
  Interventions: Procedure: Surgical Wound Infiltration

INTERVENTIONS:
Procedure: Thoracic Paravertebral Block — Thoracic paravertebral block at T3 level with bupivacaine 0.5%, dosis 1.5mg/Kg
  Arms: Thoracic Paravertebral Block
Procedure: Surgical Wound Infiltration — Surgical wound infiltration on the skin and subcutaneous tissue in surgical area with bipivacaine 0.5%, dosis 1.5mg/kg
  Arms: Surgical Wound Infiltration

SUMMARY:
Surgical treatment of breast cancer is frequently associated with postoperative pain in the surgical area. Persistent pain after breast cancer management has considerable negative effects on the quality of life of survivors. The aim of this trials is to evaluate the efficacy of thoracic paravertebral block with bupivacine 0.5% in reducing the acute pain postmastectomy compare with surgical wound infiltration with bupivacaine 0.5%.

DETAILED DESCRIPTION:
Surgical treatment of breast cancer is frequently associated with postoperative pain in the surgical area, restricted movement of the ipsilateral upper limb and increased risk of chronic pain. This usually occurs even though management with analgesics commonly used in the postoperative period. Properly treatment of acute postoperative pain have essential implications: improving the general welfare of patients, can better withstand future medical interventions, facilitating recovery in the short and long term and is believed to have positive impact on survival from cancer.

Persistent pain after breast cancer management has considerable negative effects on the quality of life of survivors. Several risks factors have been described in preoperative, intra-operative and postoperative periods of persistent or chronic pain. In the postoperative period the most important risk factor is the severity of acute pain. For this, pain relief is an essential component of care of patients undergoing breast cancer surgery. Current evidence suggests that treatment of acute postoperative pain reduces the risk of persistent or chronic pain syndrome. The surgical wound infiltration with local anesthesia has been used routinely in patients managed at the Cancer Institute and Clinica Las Americas and is described as a safe and accessible procedure for the management of acute postoperative pain. Paravertebral block represents an interesting alternative in the management of perioperative pain, often used for breast surgery, hernia repair and thoracotomy in children and adults. Although complications associated with blocking are uncommon, the implementation of Ultrasound-guided approach has become the standard for performing said method.

Such considerations have led us to evaluate whether patients with breast cancer who are undergoing mastectomy, thoracic paravertebral block could be better in relief acute pain in comparison with surgical wound infiltration with local anesthesia. This will be studied by controlled randomized to one of two intervention groups (paravertebral block or local anesthesia with infiltration of the surgical wound) allocation trial. In all patients, general anesthesia and routine postoperative analgesic is used.

ELIGIBILITY:
Inclusion Criteria:

1. Women older than 18 years.
2. Diagnosis of breast cancer requiring major elective surgery: unilateral mastectomy with or without axillary dissection; with or without axillary sentinel node biopsy; with or without immediate breast reconstruction.
3. Willingness to participate in the study during the follow-up period.

Exclusion Criteria:

1. Metastatic breast carcinoma; tumor involvement of contra lateral breast or armpit determined by clinical or paraclinical studies.
2. Medical History of coagulopathy.
3. Consumption of anticoagulants.
4. Contraindication to NSAIDs or opioids.
5. Allergy to local anesthetics of amide type.
6. Infection a interventions sites (paravertebral block or area affected breast surgical wound)
7. Pregnancy and lactation.
8. BMI>35.
9. Parkinson's disease, Alzheimer's disease or other diseases that affect the mental or motor sphere.
10. Double mastectomy or mastectomy history of previous ipsilateral to the current episode.
11. Preoperative risk classification ASA IV-V.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Acute post-surgical pain at rest and motion | 24 hours
  Acute pain at rest and in motion at 2, 4, 6, 12 and 24 hours post operative, measured by a visual analog scale (0-100 mm) for the paravertebral block group compared with the surgical wound infiltration group.

SECONDARY OUTCOMES:
Adverse Events | 2 months
  Compare the frequency and severity of adverse events in both groups
Total doses of opioids | 24 hours
  Compare the total dose of self-administered opioids analgesics for the first 24 hours
Time to the first dose of opioids | 24 hours
  Compare the time to first dose of opioids analgesics in both groups
Post-mastectomy pain syndrome | 2 months
  Compare the frequency of diagnosis of Post-mastectomy pain syndrome (SDP) two months after breast surgery in both groups
Quality of life | 2 months
  Estimate the changes in the quality of life of patients after two months after breast surgery in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Herazo, MD, MSc, Principal Investigator — Instituto de Cancerología IDC Las Américas; Hector I García, MD, MPH, MSc, Principal Investigator — Instituto de Cancerología IDC Las Américas; Jorge A Egurrola, MD, Principal Investigator — Instituto de Cancerología IDC Las Américas
Locations (1):
- Instituto de Cancerología IDC Las Américas, Medellín, Antioquia, Colombia

REFERENCES:
- [Result] Kairaluoma PM, Bachmann MS, Korpinen AK, Rosenberg PH, Pere PJ. Single-injection paravertebral block before general anesthesia enhances analgesia after breast cancer surgery with and without associated lymph node biopsy. Anesth Analg. 2004 Dec;99(6):1837-1843. doi: 10.1213/01.ANE.0000136775.15566.87. PMID 15562083
- [Result] Sidiropoulou T, Buonomo O, Fabbi E, Silvi MB, Kostopanagiotou G, Sabato AF, Dauri M. A prospective comparison of continuous wound infiltration with ropivacaine versus single-injection paravertebral block after modified radical mastectomy. Anesth Analg. 2008 Mar;106(3):997-1001, table of contents. doi: 10.1213/ane.0b013e31816152da. PMID 18292452